CLINICAL TRIAL: NCT00620360
Title: Acute Effect of Fructose on Lipid Metabolism and Gender Differences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, Professor of physiology, University of Lausanne
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 279/07/CE/FBM
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Lipid Metabolism
Keywords: dietary fructose; plasma lipids; healthy humans; gender differences; hepatic de novo lipogenesis
MeSH Terms: interventions — Fructose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fructose (Experimental): acute fructose administration
  Interventions: Dietary Supplement: fructose

INTERVENTIONS:
Dietary Supplement: fructose — acute administration of 4 times 0.3g fructose/kg lean body mass
Dietary Supplement: Fructose — acute administration of 4 times 0.3 g/kg fat-free mass oral fructose

SUMMARY:
It has been widely documented that fructose overfeeding increases plasma triglycerides and hepatic de novo lipogenesis, and impairs insulin sensitivity in healthy male volunteers. The effect of gender on the metabolic responses to fructose remains an important open question, however.

The objective of this study is to compare the effect of an acute oral fructose load on carbohydrate and lipid metabolism in healthy young males and females.

DETAILED DESCRIPTION:
The study is aimed at comparing the effects of oral fructose on several specific metabolic pathways in males and females.Participants will receive an isoenergetic diet containing 55% carbohydrate, 15% protein and 35% lipids for three days prior to testing. After this period of controlled diet, they will be studied for 2 hours in the post-absorptive state (Time 0-120 min) and over a 6 hours period (Time 120-480 min) during which they will receive 4 loads of 0,30 g/kg fat free mass U-13C labelled fructose, at times 120, 180, 240, 300. Throughout the study, deuterated glucose and glycerol will be infused to monitor whole body glucose production and glycerol turnover.

The following parameters will be monitored in basal conditions and after the ingestion of the load of fructose:

* Glycerol turnover(glycerol 2H5)
* de novo lipogenesis (incorporation of 13C into palmitate of VLDLs)
* whole body energy expenditure and net substrate oxydation (indirect calorimetry)
* net fructose oxidation (breath 13CO2)
* glucose turnover: (6,6 2H2 Glucose)
* plasma glucose, free fatty acids, ketone bodies, lactate, insulin, triacylglycerol, total cholesterol, VLDL, LDL, and HDL subfractions

An adipose tissue (periumbilical subcutaneous) biopsy will be obtaine by needle aspiration under local anesthesia in fasting conditions (time 0 min) and after fructose (time 480 min) to assess the effects of fructose on adipose gene expression profile. Key genes involved in the regulation of carbohydrate (GLUT 4, hexokinase, PDH-kinase), lipid (FAT-CD36, FABP, acetylCoA carboxylase, malonyl-CoA decarboxylase, PPARg) and energy metabolism (PGC-1a, UCP2)will be monitored

Results obtained in males and females will be compared with two-way analysis of variance

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 18-35
* Healthy
* Body mass indexes (BMI) between 19 and 25 kg/m2
* Informed consent obtained

Exclusion Criteria:

* Smokers
* Alcohol intake > 30g/day
* Drug abuse
* Diabetes mellitus

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Hepatic de novo lipogenesis | acute effect of dietary fructose (within 6 hours)

SECONDARY OUTCOMES:
Whole body lipid oxidation, glucose turnover, glycerol turnover, plasma substrates, hormone and energy expenditure (free fatty acid, glucose, lactate, beta-hydroxybutyrate, glycerol, VLDL- Triglycerides and insulin) expression of key adipose genes | acute effect of fructose (within 6 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Luc Tappy, MD, Principal Investigator — University of Lausanne
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland